CLINICAL TRIAL: NCT05434754
Title: Keeping in Touch (KiT) With Youth as They Transition to Adult Type 1 Diabetes Care: a Randomized Control Trial Testing the Effectiveness of an eHealth Text Message-based Intervention to Improve Diabetes Self-efficacy
Brief Title: Keeping in Touch (KiT) With Youth as They Transition to Adult Type 1 Diabetes Care
Acronym: KiT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Trillium Health Partners (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Rayzel Shulman, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3986
Record Dates: First submitted 2022-05-29; First posted 2022-06-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth Tool (Experimental): The Intervention is a text messaging algorithm that will operate like a chatbot, querying adolescents with T1D about their confidence with different aspects of T1D self-management as they are preparing to transition to adult diabetes care. The intervention has 4 components of messaging: personalized Educational Content, Standard Educational Curriculum, Provide participant compensation for filling out the questionnaires, Question & Answer feature.
  Interventions: Other: eHealth Tool
- Control (No Intervention): Participants randomized to the control arm will also be offered the same incentives to complete questionnaires (outcome measures) but will not receive any other components of the intervention - no personalized/customized support or diabetes resource messages and no reminders. Control arm participants will continue with their usual T1D transition care.

INTERVENTIONS:
Other: eHealth Tool — text messaging algorithm
  Arms: eHealth Tool

SUMMARY:
The investigators are testing the effectiveness of an eHealth digital tool co-designed with patients and providers to improve diabetes self-efficacy in young adults as they transition to adult type 1 diabetes care.

DETAILED DESCRIPTION:
The intervention is an eHealth digital solution co-designed with patients and providers. The intervention is a text message based algorithm that operates similar to a chatbot and will send SMS messages to participants in the experimental arm, consisting of T1D personalized support, education, resources, and a collection of outcome measures. Participants in the control arm will also be onboarded to the KiT algorithm but will only receive text-messages asking them to complete outcome measures at baseline, 6 and 12 months -- all outcome measures will be URL linkouts to REDCap surveys, housed on the SickKids REDCap servers. An embedded process evaluation of high and low engagers will also be conducted to understand how and why the intervention achieved or failed to achieve the desired effects.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 1 diabetes, ascertained from patient's medical chart
2. Receiving out-patient care for T1D at a pediatric diabetes center participating in this study
3. Is within 6 months of either planned transfer or 18th birthday so research coordinator can approach patient and inform them about the study, and then can be re-approached for consenting and enrollment only within 3-4 months of either: planned transfer to adult diabetes care OR 18th birthday
4. Proficient in written and spoken English or French
5. Possession of their own personal mobile device that can support SMS with sufficient capacity to send and receive SMS/texts
6. Valid and working mobile phone number
7. Valid email address
8. Willing to engage with intervention if randomized to intervention arm
9. Willing to complete study outcome measures (questionnaires) at all study time-points regardless of which arm they are randomized to: baseline, 6 months, and 12 months
10. Willing to provide informed consent

Exclusion Criteria:

1. Unable to carry out their diabetes care independently due to an intellectual or neurocognitive disability; discerned from medical chart during pre-screening
2. Non-resident of Ontario or Quebec
3. Planning to move out of either province in the next 6-12 months and after moving, will not be receiving diabetes care in either province and/or will not have a valid and working mobile number
4. Currently enrolled in any other clinical research trial with an SMS-based intervention
5. Currently enrolled in another diabetes intervention trial that will continue beyond the final pediatric diabetes visit

Ages: 17 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 234 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To test the effect of a text message-based T1D transition intervention compared to control at 12 months in the Self-Efficacy for Diabetes management scale. A higher score indicates better self-efficacy. | 12 months
  The primary objective of this study is to compare the effectiveness of a text message-based T1D transition intervention that will personalize transition education and support, as an adjunct to usual T1D transition care versus usual transition care alone on a patient-reported outcome measure (PROM) called the Self-Efficacy for Diabetes Management (SEDM) scale, measured at 12 months after enrollment in the study. The SEDM has scale from 1-10 where 1 denotes 'not at all sure' and 10 denotes 'completely sure' where higher scores mean better outcomes. Minimal clinically important difference is 10%.

SECONDARY OUTCOMES:
Compare text message-based T1D transition intervention to control at 6 months in the Self-Efficacy for Diabetes management scale. Higher score indicates better self efficacy. | 6 months
  A secondary objective of this study is to compare the effectiveness of a text message-based T1D transition intervention that will personalize transition education and support, as an adjunct to usual T1D transition care versus usual transition care alone on a patient-reported outcome measures (PROM) called the Self-Efficacy for Diabetes Management (SEDM) scale, measured at 6 months.
  The SEDM has scale from 1-10 where 1 denotes 'not at all sure' and 10 denotes 'completely sure' where higher scores mean better outcomes.
  Minimal clinically important difference is 10%.
To compare diabetes self-efficacy in the intervention vs. control group at baseline. A higher score indicates better self efficacy. | Baseline
  The Self-Efficacy for Diabetes Management (SEDM) scale will be used to measure diabetes self-efficacy at baseline. The SEDM has scale from 1-10 where 1 denotes 'not at all sure' and 10 denotes 'completely sure' where higher scores mean better outcomes.
  Minimal clinically important difference is 10%.
Evaluate the impact of this text message-based intervention compared to usual care at 12 months using the Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY) Tool. Higher scores indicating more confidence | 12 months
  • transition readiness measured by the Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY) tool at 12 months; READDY is a transition readiness assessment for emerging adults with diabetes diagnosed in youth. The READDY tool assesses diabetes-related knowledge or skill items by querying respondents on 42 total items split into 5 domains: knowledge, navigation, health behaviors, and insulin pump skills. Respondents answer on a Likert scale from "yes, I can do this" scored 5 to "Haven't thought about it" scored 1; confidence level is evaluated in each domain with a higher score indicating more confidence
Evaluate the impact of this text message-based intervention compared to usual care at 6 months using the Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY) Tool. Higher scores indicating more confidence | 6 months
  • transition readiness measured by the Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY) tool at 6 months; READDY is a transition readiness assessment for emerging adults with diabetes diagnosed in youth. The READDY tool assesses diabetes-related knowledge or skill items by querying respondents on 42 total items split into 5 domains: knowledge, navigation, health behaviors, and insulin pump skills. Respondents answer on a Likert scale from "yes, I can do this" scored 5 to "Haven't thought about it" scored 1; confidence level is evaluated in each domain with a higher score indicating more confidence
To compare transition readiness in the intervention and control groups at baseline using the Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY) Tool. Higher scores indicating more confidence | Baseline
  • transition readiness measured by the Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY) tool at baseline. READDY is a transition readiness assessment for emerging adults with diabetes diagnosed in youth. The READDY tool assesses diabetes-related knowledge or skill items by querying respondents on 42 total items split into 5 domains: knowledge, navigation, health behaviors, and insulin pump skills. Respondents answer on a Likert scale from "yes, I can do this" scored 5 to "Haven't thought about it" scored 1; confidence level is evaluated in each domain with a higher score indicating more confidence
Evaluate the impact of this text message-based intervention compared to usual care at 12 months on self-reported Barriers to Diabetes Adherence in Adolescence questionnaire (BDA) Stigma subscale | 12 months
  • perceived stigma of living with T1D using the Barriers to Diabetes Adherence in Adolescence questionnaire (BDA) Stigma Subscale; in our study, stigma will be defined as an affirmative response to at least one of three key items on this subscale. The scale ranges from "not at all true" (1) to "completely true" (5). Where a score greater than 2 to at least 1 of 3 key items indicates stigma.
Evaluate the impact of this text message-based intervention compared to usual care at 6 months on self-reported Barriers to Diabetes Adherence in Adolescence questionnaire (BDA) Stigma subscale | 6 months
  • perceived stigma of living with T1D using the Barriers to Diabetes Adherence in Adolescence questionnaire (BDA) Stigma Subscale; in our study, stigma will be defined as an affirmative response to at least one of three key items on this subscale. The scale ranges from "not at all true" (1) to "completely true" (5). Where a score greater than 2 to at least 1 of 3 key items indicates stigma.
To compared perceived stigma of living with T1D between the intervention and control groups at baseline using the self-reported Barriers to Diabetes Adherence in Adolescence questionnaire (BDA) Stigma subscale | baseline
  • perceived stigma of living with T1D using the Barriers to Diabetes Adherence in Adolescence questionnaire (BDA) Stigma Subscale; in our study, stigma will be defined as an affirmative response to at least one of three key items on this subscale. The scale ranges from "not at all true" (1) to "completely true" (5). Where a score greater than 2 to at least 1 of 3 key items indicates stigma.
Evaluate the impact of this text message-based intervention compared to usual care at 12 months using self-reported A1c values | 12 months
  • A1c will be self-reported in the following categories of values: < 7%, 7 to < 8%, 8 to < 9%, >9% where higher percentage indicates poorer diabetes management
Evaluate the impact of this text message-based intervention compared to usual care at 6 months using self-reported A1c | 6 months
  A1c will be self-reported in the following categories of values: < 7%, 7 to < 8%, 8 to < 9%, >9% where higher percentage indicates poorer diabetes management
To compare A1c between the intervention and control groups at baseline by measuring self-reported A1c | baseline
  A1c will be self-reported in the following categories of values: < 7%, 7 to < 8%, 8 to < 9%, >9% where higher percentage indicates poorer diabetes management
Evaluate the impact of this text message-based intervention compared to usual care on number of diabetes-related ED visits during the 12 months of intervention | 12 months
  • Health administrative data from ICES in Ontario and RAMQ in Quebec will be collected during the 12 months of intervention. ICES is an independent, not-for-profit research institute made up of a community of research, data and clinical experts in Ontario. RAMQ manages, administers and publishes health data in the province of Quebec.
To compare the number of diabetes-related ED visits in the 24 months prior to enrolment in the intervention vs. control group at baseline | baseline
  • Health administrative data from ICES in Ontario and RAMQ in Quebec will be collected during the 24 months prior to enrolment. ICES is an independent, not-for-profit research institute made up of a community of research, data and clinical experts in Ontario. RAMQ manages, administers and publishes health data in the province of Quebec.
Evaluate the impact of this text message-based intervention compared to usual care on number of diabetes-related hospitalizations and length of diabetes-related hospitalizations during the 12 months of intervention | 12 months
  • Health administrative data from ICES in Ontario and RAMQ in Quebec will be collected during the 12 months of intervention. ICES is an independent, not-for-profit research institute made up of a community of research, data and clinical experts in Ontario. RAMQ manages, administers and publishes health data in the province of Quebec.
Number of diabetes-related hospitalizations and length of diabetes-related hospitalizations 24 months prior to intervention for both intervention and control populations to describe baseline characteristics | Baseline
  • Health administrative data from ICES in Ontario and RAMQ in Quebec will be collected during the 24 months prior to enrolment. ICES is an independent, not-for-profit research institute made up of a community of research, data and clinical experts in Ontario. RAMQ manages, administers and publishes health data in the province of Quebec.
Evaluate the impact of this text message-based intervention costs compared to usual care costs | 12 months
  * Costs of implementation will be collected to ascertain the cost of developing and using this intervention in a hospital setting in Ontario and Quebec; variables that will be collected for this analysis will include: salaries for staff working on the design, development and management of the intervention for the entire intervention duration; salary of research coordinators working to onboard participants to the intervention; cost of digital services and office equipment needed to develop and manage the intervention (computers, hosting service, servers); cost of REDcap servers and hospital IT support for REDCap integration with MEMOTEXT platform
  * Aggregate and direct medical costs associated with the intervention and its implementation will be measured for the 12 months of the intervention duration using study and administrative data
Exploring how the KiT large language model (LLM) chatbot is used in a real-world setting. | 12 months
  * Analyses for the preliminary safety and performance KiT LLM chatbot testing will include descriptively describing whether the LLM Evaluator acts more conservatively than human raters when scoring answers, and if the answers generated by KiT LLM are acceptable based on the graded criteria.
  * After the trial is completed, the investigators will analyze conversation logs between participants and KiT LLM to derive effective engagement with the bot. This will include analyzing the conversation between participants and KiT LLM (eg, duration, breadth, and depth of bot usage).
  * The performance of the LLM Evaluator will also be assessed by evaluating conversations flagged and any potentially sensitive conversations missed. This evaluation will provide insights into how KiT LLM was used in a real-world setting and opportunities to improve its performance over time.

OTHER OUTCOMES:
Evaluation of participant engagement with the intervention with number of participants who are engaging with intervention messages | 12 months
  Embedded process evaluation using real-time engagement metrics with number of participants who are engaging with intervention messages on Concurrent process evaluation allows for real-time intervention modification to increase and improve user engagement and content delivery
Evaluation of participant engagement with the intervention looking at which types of messages are the most and least engaged with | 12 months
  Embedded process evaluation using real-time engagement metrics looking at which types of messages are the most and least engaged with Concurrent process evaluation allows for real-time intervention modification to increase and improve user engagement and content delivery
Evaluation of intervention fidelity | 12 months
  Embedded process evaluation using real-time engagement metrics (i.e. number of participants who are engaging with intervention messages on and which types of messages are the most and least engaged with) Concurrent process evaluation allows for real-time intervention modification to increase and improve user engagement and content delivery
Identify the different paths of engagement (i.e., combinations of KiT components) that produce a positive effect on trial outcomes). Specifically from when the chatbot was incorporated in September 2024. | 12 months.
  The investigators will identify the potential paths and corresponding combination of factors that are associated with trial outcomes using Coincidence Analysis.

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Oak Valley Health, Markham, Ontario
  - Trillium Health Partners, Mississauga, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
  - Saint Justine Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanmugalingham G, Mok E, Cafazzo JA, Desveaux L, Brazeau AS, Booth GL, Greenberg M, Kichler J, Rac VE, Austin P, Goldbloom E, Henderson M, Landry A, Zenlea I, Taylor M, Nakhla M, Shulman R. Text message-based intervention, Keeping in Touch (KiT), to support youth as they transition to adult type 1 diabetes care: a protocol for a multisite randomised controlled superiority trial. BMJ Open. 2023 May 8;13(5):e071396. doi: 10.1136/bmjopen-2022-071396. PMID 37156577

DOCUMENTS (1):
  • Study Protocol (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT05434754/Prot_001.pdf